CLINICAL TRIAL: NCT00162968
Title: Escitalopram as a Treatment for Pain in Polyneuropathy. A Double-Blind, Randomized, Placebo Controlled Trial.
Brief Title: Escitalopram as a Treatment for Pain in Polyneuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); H. Lundbeck A/S (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: escit01
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Pain; Polyneuropathies
Keywords: polyneuropathies; pain; drug effects; escitalopram; serotonin uptake inhibitors
MeSH Terms: conditions — Pain; Polyneuropathies | interventions — Escitalopram

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
Many people with polyneuropathy suffer from pain which is difficult to treat. Escitalopram is a relatively new drug used in the treatment of depression. Escitalopram's action mechanism on the brain suggests that escitalopram also may have an effect on neuropathic pain. This study will test the efficacy of escitalopram in patients with painful polyneuropathy.

DETAILED DESCRIPTION:
Tricyclic antidepressants appear to be the most efficacious treatment of painful polyneuropathy. However, these drugs are contraindicated in some patients and a substantial number of patients decline treatment due to side-effects. Therefore, effective drugs that are better tolerated are needed. Clinical and basic research has demonstrated that drugs with serotonergic action can alleviate neuropathic pain. Escitalopram increases serotonin concentration in the central nervous system, suggesting that it might be a potential alternative to current treatments of neuropathic pain. The aim of this study is to test if escitalopram would relieve painful polyneuropathy.

Comparisons: Treatment with 20 mg escitalopram daily will be compared in a cross-over design with placebo. Each treatment period will last 6 weeks. During the last week of each treatment period, the dose will be tapered.

ELIGIBILITY:
Inclusion Criteria:

* median total pain score at baseline week >=4 on a 10 point numerical rating scale
* characteristic symptoms of polyneuropathy within at least 6 months
* diagnosis confirmed by physical examination, neurophysiologic exam. and/or quantitative sensory testing
* pain at least 4 of 7 days
* fertile women are using anticonceptive

Exclusion Criteria:

* other cause to pain than polyneuropathy
* former allergic reactions on escitalopram
* known adverse events on escitalopram
* pregnancy or nursing
* critical disease (terminal cancer, cardial incompensation or critical renal or lung disease)
* treatment with monoamine oxidase inhibitors between the trial or 2 weeks before or after treatment with other antidepressants, antiepileptic agents or opioids

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-12; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
pain relief

SECONDARY OUTCOMES:
effect on total pain and different subtypes of pain
effect on quantitative sensory testing
effect on pain related sleep disturbances
effect on quality of life
to determine if depression before treatment predicts an eventual pain relieving effect of escitalopram

CONTACTS AND LOCATIONS:
Overall Officials: Soeren H Sindrup, MD, PhD, Principal Investigator — Odense University Hospital, Dept. of neurology
Locations (2):
- Denmark (2):
  - Danish Pain Research Center, Aarhus University Hospital, Noerrebrogade 44, Aarhus
  - Dept. of Neurology, Odense University Hospital, Sdr. Boulevard 29, Odense

REFERENCES:
- [Background] Burke WJ. Escitalopram. Expert Opin Investig Drugs. 2002 Oct;11(10):1477-86. doi: 10.1517/13543784.11.10.1477. PMID 12387707
- [Background] Sindrup SH, Jensen TS. Pharmacologic treatment of pain in polyneuropathy. Neurology. 2000 Oct 10;55(7):915-20. doi: 10.1212/wnl.55.7.915. PMID 11061244
- [Background] Woolf CJ, Mannion RJ. Neuropathic pain: aetiology, symptoms, mechanisms, and management. Lancet. 1999 Jun 5;353(9168):1959-64. doi: 10.1016/S0140-6736(99)01307-0. PMID 10371588
- [Background] Mork A, Kreilgaard M, Sanchez C. The R-enantiomer of citalopram counteracts escitalopram-induced increase in extracellular 5-HT in the frontal cortex of freely moving rats. Neuropharmacology. 2003 Aug;45(2):167-73. doi: 10.1016/s0028-3908(03)00138-2. PMID 12842122